CLINICAL TRIAL: NCT06985147
Title: A Phase 2, Open-Label Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of DISC-3405 in Participants With Polycythemia Vera (PV)
Brief Title: A Phase 2, Open-Label Study of DISC-3405 in Participants With Polycythemia Vera (PV)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DISC-3405-201
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Polycythemia Vera (PV)
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: Up to 3 cohorts of participants are planned:
  * Cohort A will include 20 participants. The first 4 participants enrolled will be administered a starting dose level of Dose A DISC-3405 subcutaneous which will be followed by within-participant dose escalation. Following Safety Review Committee review of the data, an additional 16 participants will be enrolled and administered a starting dose level of Dose B DISC-3405 subcutaneous.
  * Cohort B will enroll up to 20 participants administered a dose level of Dose B DISC-3405 subcutaneous once every 4 weeks.
  * Cohort C is optional and will enroll up to 20 participants administered a dose level up to that previously studied of DISC-3405 subcutaneous once every 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Within-participant dose escalation (Experimental): This is an open-label, multicenter, within-participant dose escalation study examining up to 2 dose levels of DISC-3405.
  Interventions: Drug: DISC-3405

INTERVENTIONS:
Drug: DISC-3405 — DISC-3405 is administered subcutaneously.

SUMMARY:
This open-label, multicenter, within-participant dose escalation study examining up to 2 dose levels of DISC-3405 will assess the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of DISC-3405 in participants with polycythemia vera (PV).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of signing the informed consent form (ICF).
2. Meet revised 2022 World Health Organization (WHO) criteria for the diagnosis of PV.
3. Complete blood count values at Screening of HCT <45% or HCT <48% if followed by a phlebotomy within 2 weeks, white blood cells 4000/μL to 20,000/μL (inclusive), and platelets 100,000/μL to 1,000,000/μL (inclusive).
4. At least 3 phlebotomies in 26 weeks before Screening or at least 5 phlebotomies in 52 weeks before Screening. At least 1 phlebotomy must be within the 12 weeks prior to Screening.
5. Participants receiving cytoreductive therapy must have been taking for at least 6 months and be on a stable PV therapy regimen for at least 2 months for hydroxyurea, interferon or ruxolitinib with no anticipated need for dose adjustments during the study, or have decreasing dose (with medical monitor approval).
6. Participants treated with phlebotomy alone must have stopped cytoreductive therapy 6 months before Screening.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, or with medical monitor approval, ECOG 2.
8. If male with female sexual partner(s) of childbearing potential, agrees to use one of the following acceptable methods of contraception during the study and for at least 120 days after the last study drug dose:

   1. Stable hormonal contraceptive (≥3 months; female partner) in conjunction with a barrier method (eg, condom or diaphragm [female partner])
   2. Intrauterine device in place for at least 3 months (female partner)
   3. Surgically sterile hysterectomy, bilateral oophorectomy, or bilateral tubal ligation (female partner) in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
   4. Confirmed successful vasectomy in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
9. If female, then EITHER postmenopausal, defined as at least 12 months of natural, spontaneous amenorrhea, 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone >40 mIU/mL at Screening, or at least 6 weeks following surgical menopause (bilateral oophorectomy with or without hysterectomy); surgically sterile, OR agreeable to use of highly effective contraception (listed below) on Day 1 (or earlier) and for at least 120 days after the last dose of study drug:

   1. Stable hormonal contraceptive (≥3 months) in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
   2. Intrauterine device in place for at least 3 months
   3. Tubal ligation or single male partner with vasectomy in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
10. Negative pregnancy test (females of childbearing potential).
11. Able to understand the study aims, procedures, and requirements, and provide written informed consent.
12. Able to comply with all study procedures.

Exclusion Criteria:

1. Clinically significant laboratory abnormalities at Screening.
2. Participants who require phlebotomy at HCT levels <45%.
3. Clinically significant thrombosis (eg, deep vein thrombosis or splenic vein thrombosis) within 2 months prior to study treatment.
4. Clinically significant active or chronic bleeding, considered meaningful in consultation with the medical monitor, within 6 months prior to study treatment.
5. Significant renal dysfunction, evidenced by estimated glomerular filtration rate of <30 mL/min/1.73 m2 at the Screening visit, as assessed locally.
6. History of invasive malignancies within the last 5 years, except localized cured prostate cancer and cervical cancer, or other malignancies deemed acceptable by the Sponsor.
7. Participants with in situ or stage 1 squamous cell carcinoma of the skin, in situ or stage 1 basal cell carcinoma of the skin, or in situ melanoma of the skin identified during Screening unless the cancer is adequately treated before study entry.
8. Received busulfan, pipobroman, or phosphorus-32 within 7 months prior to Screening.
9. Major surgery within 8 weeks before Screening or incomplete recovery from any previous surgery.
10. A history or known allergic reaction to any investigational product excipients or history of anaphylaxis to any food or drug.
11. History of alcohol dependence or excessive alcohol consumption, as assessed by the Investigator.
12. Active human immunodeficiency virus (HIV), hepatitis B or C. A positive hepatitis or HIV result should be discussed between the Investigator and Sponsor prior to enrollment.
13. Other medical or psychiatric condition or laboratory finding not specifically noted above that, in the judgment of the Investigator or Sponsor, would put the participant at unacceptable risk or otherwise preclude the participant from participating in the study.
14. Condition or concomitant medication that would confound the ability to interpret clinical data, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months.
15. If female, pregnant or breastfeeding.
16. Participation in any other clinical protocol or investigational study that involves administration of experimental therapy and/or therapeutic devices within 30 days (or 5 half-lives for drugs, whichever is longer) of Screening. Previous use of other hepcidin inducing agents that may impact TMPRSS6 expression are not allowed. Previous use of hepcidin mimetics may be allowed in discussion with the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | Up to 365 days
  Proportion of participants with treatment-emergent adverse events
Incidence of clinically abnormal vital signs | Up to 365 days
  Proportion of participants with changes in vital signs
Incidence of clinically abnormal physical exam | Up to 365 days
  Proportion of participants with changes in physical examinations
Incidence of clinically abnormal electrocardiograms | Up to 365 days
  Proportion of participants with changes in electrocardiograms (ECGs)
Incidence of abnormal laboratory test results | Up to 365 days
  Proportion of participants with changes in clinical laboratory results

SECONDARY OUTCOMES:
Proportion of participants achieving therapeutic response, defined as absence of phlebotomy eligibility, during the maintenance period | Up to 365 days
Number of phlebotomies during the maintenance and optimization periods | Up to 365 days
Proportion of participants achieving therapeutic response, defined as absence of phlebotomy eligibility, during the optimization period | Up to 365 days
Proportion of participants with HCT values <45% throughout the study | Up to 365 days
Area under the plasma concentration versus time curve (AUC) following the first dose | Up to 365 days
Peak plasma concentration (Cmax) following the first dose | Up to 365 days
Elimination half-life (t½el) following the first dose | Up to 365 days
Apparent clearance (CL/F) following the first dose | Up to 365 days
Maximum concentration at steady state (Cmax_ss) after repeating doses | Up to 365 days
Pre-dose trough concentration (Ctrough) after repeating doses | Up to 365 days
Change from baseline for HCT | Up to 365 days
Change from baseline for serum hepcidin-25 | Up to 365 days
Change from baseline for serum iron | Up to 365 days
Apparent volume of distribution (Vd/F) | Up to 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD PhD, Study Director — Disc Medicine
Locations (11):
- United States (11):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - UCLA Health, Los Angeles, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Minnesota, Rochester, Minnesota
  - Siteman Cancer Center - Washington University St. Louis, St Louis, Missouri
  - Atrium Health - Levine Cancer Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No